CLINICAL TRIAL: NCT04975035
Title: A Prospective, Open-ended, Multi-center Study of Schizophrenia Patients Switching to Zolodine
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-074
Record Dates: First submitted 2021-06-20; First posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2012-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

ARMS (1):
- Zolodine group (Experimental)
  Interventions: Drug: Zolodine

INTERVENTIONS:
Drug: Zolodine — Collect 200 patients who meet the criteria into the group. After enrollment, according to the principle of cross dressing change, the attending physician can decide the dressing change method according to the patient's condition, individual condition and other factors; within 2-4 weeks, the original antipsychotics should be gradually stopped, and Zoladine capsules will be gradually added to the target The dose is 120-160mg/d, orally 1-2 times a day, with meals.

SUMMARY:
Through self-controlled studies on metabolic syndrome related indicators, efficacy and other adverse reactions in patients with schizophrenia who developed metabolic syndrome after treatment with other antipsychotics, switched to Zoladine capsules (ziprasidone hydrochloride capsules). To evaluate the clinical application value of switching to Zolodine for schizophrenia patients with metabolic syndrome, and to explore the drug selection strategy for long-term treatment of schizophrenia patients.

ELIGIBILITY:
Inclusion Criteria:

* Meet the DSM-IV diagnostic criteria for schizophrenia, patients aged 18-40 years old have been treated with other antipsychotics for more than 8 weeks (inclusive) before being included, meet the diagnostic criteria for metabolic syndrome (IDF, 2005), and have not reached diabetes , Patients with diagnostic criteria for hypertension.

Exclusion Criteria:

* Female patients who are pregnant or breastfeeding;
* Serious and unstable physical diseases, including: cardiovascular, respiratory, liver, kidney, gastrointestinal, nerve, endocrine, immune, blood system, narrow-angle glaucoma, history of seizures;
* Patients with refractory schizophrenia;
* Those who meet the DSM-IV standards for dementia or substance dependence (except tobacco);
* Patients with a history of contraindications to ziprasidone or intolerance of ziprasidone;
* Patients who use long-acting antipsychotic injections or oral medications;
* Patients who have recently experienced prolonged QT interval, acute myocardial infarction, and decompensated heart failure;
* Patients have recently taken drugs that can prolong the QT interval, such as dofetilide, sotalol, quinidine, other class Ia and III antiarrhythmic drugs, mesoridazine, thioridazine, Chlorpromazine, droperidol, pimozide, sparfloxacin, gatifloxacin, moxifloxacin, halofantrine, mefloquine, pentamidine, arsenic trioxide, levomethadone, dolastron methanesulfonate Acid, probucol or tacrolimus;
* At the same time taking other drugs that can cause obesity, such as oral contraceptives;
* Patients who have met metabolic syndrome before diagnosis and treatment of schizophrenia.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2012-01-01; Primary Completion 2012-07-01 (Actual); Study Completion 2012-07-01 (Actual)

PRIMARY OUTCOMES:
score of PANSS | 2 weeks
  the score of positive and negative syndrome scale (PANSS), the minimum and maximum values are 16 and 112, the higher scores mean a worse outcome.
score of HAMA | 2 weeks
  the score of Hamilton anxiety scale(HAMA), the minimum and maximum values are 0 and 56, the higher scores mean a worse outcome.
score of HAMD | 2 weeks
  the score of Hamilton depression scale(HAMD), the minimum and maximum values are 0 and 68, the higher scores mean a worse outcome.